CLINICAL TRIAL: NCT00079703
Title: Diet, Genetics, and CVD Risk Factor Response in Blacks
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1245; U01HL072510 (NIH)
Record Dates: First submitted 2004-03-10; First posted 2004-03-15 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To test the hypothesis that the responsiveness of major and emerging cardiovascular disease risk factors to changes in diet composition clusters within families depending on genetic susceptibility factors.

DETAILED DESCRIPTION:
BACKGROUND:

Reduction in risk of cardiovascular disease (CVD) through dietary change has considerable potential for a beneficial impact on public health. On a population basis, moderation of both lipid profiles and blood pressure can be accomplished readily with a prudent diet. Nevertheless, individual response to dietary impact on CVD risk factors varies widely, presumably as a result of genetic differences. In particular, Blacks who constitute a subpopulation with documented increased risk of morbidity and mortality from CVD would disproportionately benefit from interventions designed to maximize the impact of dietary change tailored to individual genetic makeup. Therefore, study of the influence of diet on CVD risk factors, along with enhanced understanding of the genetic components involved, would greatly potentiate chronic disease interventions.

The study is conducted in response to a Request for Applications issued in October, 2001 on the Interaction of Genes and the Environment in Shaping Risk Factors for Heart, Lung, Blood, and Sleep Disorders.

DESIGN NARRATIVE:

Two-generational family lines will be identified in Blacks with elevated low density lipoprotein-C (LDLC) in probands. The population will be fed a controlled diet contrasting an established heart healthy regimen with a typical American one. Concomitant rigorous genetic, anthropometric, and behavioral evaluation will provide data with which to analyze individual differences in response to consistent dietary intake. In Specific Aim 1, Black, two-generational, families will be recruited and provided interventional diets designed to reduce (or not) LDL-C and blood pressure. In Specific Aim 2, non-genetic predictors of CVD risk factor response will be identified through extensive assessments of baseline behavioral characteristics, anthropometric features, and metabolic factors. In Specific Aim 3, the underlying genetic factors that predispose to response (or the lack of) to dietary interventions will be identified through the examination of polymorphisms in candidate genes and the identification of susceptibility loci by linkage analyses. In Specific Aim 4, interactions between diet, CVD risk factor response and genetic factors will be dissected through measures of potential mediating metabolic pathways.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael LeFevre — LSU Pennington Biomedical Research Center

REFERENCES:
- [Derived] Law HG, Khan MA, Zhang W, Bang H, Rood J, Most M, Lefevre M, Berglund L, Enkhmaa B. Reducing saturated fat intake lowers LDL-C but increases Lp(a) levels in African Americans: the GET-READI feeding trial. J Lipid Res. 2023 Sep;64(9):100420. doi: 10.1016/j.jlr.2023.100420. Epub 2023 Jul 22. PMID 37482217